CLINICAL TRIAL: NCT01515046
Title: Pharmacological Ascorbate for the Control of Metastatic and Node-Positive Pancreatic Cancer (PACMAN): A Phase II Trial
Brief Title: Clinical Trial of High-dose Vitamin C for Advanced Pancreatic Cancer
Acronym: PACMAN-II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Standard of care changed to FOLFIRINOX; poor accrual.
Sponsor: Joseph J. Cullen (Other)
Collaborators: Susan L Bader Foundation of Hope (Unknown); Holden Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Joseph J. Cullen, Professor of Surgery, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201204737; P30CA086862 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer
Keywords: Vitamins; Complementary medicine; Pancreatic cancer; Ascorbate; Ascorbic Acid; Antioxidants; Gemcitabine; Pharmacologic actions
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine with escalating IV ascorbate (Experimental): Gemcitabine (1000 mg/m2) weekly for three weeks and then one week off. Ascorbic Gemcitabine (1000 mg/m2) weekly for three weeks and then one week off.
  Ascorbate (vitamin C) given twice weekly, escalating doses weekly. Week 1: 15 grams ascorbate / infusion for two infusions. Doses are then escalated in 25 gram increments until therapeutic window is achieved (350 mg/dL or above). Dose is then held at that level for the full cycle.
  Interventions: Drug: Gemcitabine with escalating ascorbic acid

INTERVENTIONS:
Drug: Gemcitabine with escalating ascorbic acid — Gemcitabine 1000 mg/m2 weekly for 3 weeks with one week off (this is 1 cycle)
  Ascorbate dose is targeted to achieve plasma level of 350 mg/dL. Infusions are given twice weekly, each week of a cycle (4 weeks to a cycle)
  Other Names: Gemzar; Ascorbic Acid for Infusion, USP

SUMMARY:
This is a phase II study. It is designed to provide information about if high-dose ascorbate (vitamin C) increases survival for pancreatic cancer patients. The hypothesis is that vitamin C is well tolerated and increases cancer treatment effectiveness, lengthening survival time for patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
Adenocarcinoma of the pancreas is the fourth leading cause of cancer death in the United States and is increasing in incidence; the prognosis remains dismal. We propose to investigate an entirely new approach, using pharmacological ascorbate, combined with Gemcitabine, to treat this cancer. Intravenous ascorbate (i.e., ascorbic acid, vitamin C), but not oral ascorbate, produces high plasma concentrations, which are in the range that can be cytotoxic to tumor cells. Though ascorbate has been utilized in cancer therapy, few studies have investigated intravenous deliver of ascorbate. Preliminary studies from our group have demonstrated that ascorbate induces oxidative stress and cytotoxicity in pancreatic cancer cells; this cytotoxicity appears to be greater in tumor vs. normal cells. We hypothesize that production of H2O2 mediates the increased susceptibility of pancreatic cancer cells to ascorbate-induced metabolic oxidative stress. Gemcitabine is the standard chemotherapy drug used to treat pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cytological or histological diagnosis of adenocarcinoma arising in the pancreas. Diagnosis from metastatic sampling is acceptable.
* Disease must be measured radiologically.
* Failed initial therapy or ineligible for definitive curative therapy.
* If prior treatment included radiation therapy, recurrent disease must be outside of the targeted volume.
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky > 50%, see Appendix A).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3,000/mm3
  * absolute neutrophil count ≥ 1,500/mm3
  * platelets ≥ 100,000/mm3
  * total bilirubin < 2x institutional upper limit of normal
  * AST(SGOT) < 3x institutional upper limit of normal OR < 5x institutional upper limit of normal for patients presenting with liver metastases
  * ALT (SGPT) < 3x institutional upper limit of normal OR < 5x institutional upper limit of normal for patients presenting with liver metastases
  * PT/INR within normal institutional limits, unless patient is on warfarin or other antithrombotic agents
  * creatinine < 1.5 X institutional upper limit of normal OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * Not pregnant. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy to treat metastatic disease.
* Adjuvant therapy (including radiation therapy) within 4 calendar weeks.
* Unresolved toxicities from prior therapy for the malignancy.
* G6PD (glucose-6-phosphate dehydrogenase) deficiency.
* Second malignancy other than non-melanoma skin cancers within the past 5 years.
* Excess consumption of alcohol where an excess of alcohol is defined as more than four of any one of the following per day: 30 mL distilled spirits, 340 mL beer, or 120 mL wine.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations, or any other condition that would limit compliance with study requirements as determined by study team members.
* Pregnant or lactating women: The risks of chemotherapy to a fetus/infant are well documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Cullen, MD, Principal Investigator — University of Iowa; Joseph J Cullen, MD, Study Chair — University of Iowa
Locations (1):
- The Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cullen JJ. Ascorbate induces autophagy in pancreatic cancer. Autophagy. 2010 Apr;6(3):421-2. doi: 10.4161/auto.6.3.11527. Epub 2010 Apr 15. PMID 20400857
- [Background] Du J, Martin SM, Levine M, Wagner BA, Buettner GR, Wang SH, Taghiyev AF, Du C, Knudson CM, Cullen JJ. Mechanisms of ascorbate-induced cytotoxicity in pancreatic cancer. Clin Cancer Res. 2010 Jan 15;16(2):509-20. doi: 10.1158/1078-0432.CCR-09-1713. Epub 2010 Jan 12. PMID 20068072
- [Background] Welsh JL, Wagner BA, van't Erve TJ, Zehr PS, Berg DJ, Halfdanarson TR, Yee NS, Bodeker KL, Du J, Roberts LJ 2nd, Drisko J, Levine M, Buettner GR, Cullen JJ. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol. 2013 Mar;71(3):765-75. doi: 10.1007/s00280-013-2070-8. Epub 2013 Feb 5. PMID 23381814

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine With Escalating IV Ascorbate: Gemcitabine (1000 mg/m2) weekly for three weeks and then one week off. Ascorbic Gemcitabine (1000 mg/m2) weekly for three weeks and then one week off.
  Ascorbate (vitamin C) given twice weekly, escalating doses weekly. Week 1: 15 grams ascorbate / infusion for two infusions. Doses are then escalated in 25 gram increments until therapeutic window is achieved (350 mg/dL or above). Dose is then held at that level for the full cycle.
  Gemcitabine with escalating ascorbic acid: Gemcitabine 1000 mg/m2 weekly for 3 weeks with one week off (this is 1 cycle)
  Ascorbate dose is targeted to achieve plasma level of 350 mg/dL. Infusions are given twice weekly, each week of a cycle (4 weeks to a cycle)
Period: Overall Study
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time to event outcome measure (death), measured in days from cycle 1 day 1.
Time Frame: up to 5 years
Measure: Number; unit: days
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 1
days | 268

2. Secondary Outcome: Progression Free Survival
Description: Time-to-event outcome measure (initial disease progression) measured in days from cycle 1 day 1 to day of first progression as defined by RECIST criteria from NCI.
Time Frame: up to 5 years
Measure: Number; unit: days
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 1
days | 80

3. Secondary Outcome: Number of Drug-related Adverse Events Per Cycle
Description: Adverse events linked to ascorbate will be categorized and quantified using CTCAE v4 at the bottom of each cycle. Incidence and frequency will be compared to scientific literature
Time Frame: every 28 days up to 5 years
Population: Due to n=1 and study termination, the data were not analyzed.
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 0
Value | 0

4. Secondary Outcome: F2-isoprostane Levels
Description: F2-isoprostane is a marker of systemic oxidative stress.
Time Frame: Once every 28 days for up to 5 years
Population: Due to n=1 and study termination, the data were not analyzed.
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 0

5. Secondary Outcome: Ascorbate Levels
Description: Ascorbate levels will be taken at the bottom of each cycle to assess therapeutic dose window.
Time Frame: Once every 28 days up to 5 years
Arm/Group | Gemcitabine With Escalating IV Ascorbate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Events collected over one calendar year
Description: Adverse event reporting is consistent with the definition provided by clinicaltrials.gov
Arm/Group | Gemcitabine With Escalating IV Ascorbate
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine With Escalating IV Ascorbate (N=1)
Anemia, grade 1 (Investigations) | 1 (1) — Hemoglobin, Low
white blood cell count, decreased, grade 1 (Investigations) | 1 (1) — leukopenia leukocytes, low
Lymphocyte count decreased, grade 2 (Investigations) | 1 (1) — lymphopenia
neutrophil count decreased, grade 3 (Investigations) | 1 (1) — neutropenia
platelet count decreased, grade 3 (Investigations) | 1 (1)
Alanine aminotransferase increased, grade 1 (Investigations) | 1 (1) — ALT increased SGPT increased

LIMITATIONS AND CAVEATS:
There was only one treated participant. Conclusions cannot be drawn from these data due to limited sampling size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes